CLINICAL TRIAL: NCT06089759
Title: Performance and Safety of the Lipo-transfer Cannulas in Patients Underlying Lipofilling Treatment
Status: Completed | Type: Observational
Sponsor: Aesthetic Group (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: LIPOTRANSFER
Record Dates: First submitted 2023-08-21; First posted 2023-10-18 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Lipodystrophy; Deformities
Keywords: Lipofilling; Liposuction; Fat injection; Repair and aesthetic surgery; Aesthetic body contouring
MeSH Terms: conditions — Lipodystrophy; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this post-market clinical follow up study is to assess the safety and performance of Aesthetic Group cannulas. The study will evaluate the outcome of the Aesthetic Group cannulas range over a period of 1 month after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years at intervention
* Patient who will undergo a lipofilling treatment with at least one cannula of Aesthetic Group
* Patient informed of his/her participation and willing to participate in the study.
* Patient able to read, write and understand French.

Exclusion Criteria:

* Patient deprived of freedom, under guardianship/curatorship or placed under judicial protection
* Patient unable to follow study procedures
* Patient with hematologic abnormalities, prior radiotherapy or chemotherapy
* Chronic use of medicines or drugs
* Patient with diabetes mellitus
* Patient with connective tissue diseases, any type of fat tissue disorder (lipodystrophy)
* Patient with bleeding disorders; immune deficits; heart, liver, and kidney insufficiency
* Patient with allergies to local anaesthetics
* Patient with pacemaker and serious heart rhythm disorders
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is directly linked to target population for autograft with Aesthetic group's cannulas
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The performance of the cannulas for infiltration, fat harvesting or fat injection. | D0 (at intervention)
  The success rate of cannulas defined by the capacity to infiltrate, harvest or inject.

SECONDARY OUTCOMES:
The surgeon's satisfaction with the procedure | D0 (at intervention)
  The surgeon satisfaction will be assessed using a 4-point scale (likert scale) at intervention. (Very satisfied, Satisfied, Unsatisfied, Very unsatisfied). Very satisfied is the higher score and outcome.
The safety of the cannulas during the intervention (All adverse device effects occurred during the intervention will be summarized) | D0 (at intervention)
  All adverse device effects occurred during the intervention
The safety of the intervention within the 1 month post intervention (All adverse events occurred from the intervention to the 1 month follow-up visit will be summarized) | D0 (at intervention) to month 1
  All adverse events occurred from the intervention to the 1 month follow-up visit
The usability of the cannulas during the intervention | D0 (at intervention)
  Usability of the cannulas (easy to fit, …) assessed with a questionnaire (Scale of ease of fitting the cannula) in by the investigator (Very satisfied, Satisfied, Unsatisfied, Very unsatisfied). "Very satisfied" is the best value and outcome.
The quality of life | At baseline and 1 month follow-up
  Improvement of QoL score (numeric scale, 0 to 10, 10 is the maximum and the best value, 0 is the minimum value) at 1 month compared with pre-operative visit
The patient's satisfaction at 1 month (binary variable) | At 1 month
  The proportion of patients who are satisfied at 1 month (binary variable, yes or no, yes is the best value)
The surgeon's satisfaction at 1 month | At 1 month
  The proportion of patients for whom the surgeon is satisfied at 1 month
The improvement of skin quality/aesthetic (likert scale) | At 1 month
  The proportion of patients where the skin quality/aesthetic is improved at each follow-up visit. (Good improvement, mild improvement, no improvement, worsening, "good improvement" is the best value and outcome, "worsening" is the minimum value)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique Pasteur, Brest
  - Clinique Phenicia, Marseille
  - Clinique Eiffel, Paris